CLINICAL TRIAL: NCT02467855
Title: A Multi-Centre, Non-Interventional, Hospital-Based, Cross-Sectional as Well as Longitudinal Epidemiological Study in Thai Subjects With Hypertension
Brief Title: Epidemiological Study in Thai Participants With Hypertension
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: AZI-P4-003
Record Dates: First submitted 2015-04-23; First posted 2015-06-10 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
Keywords: Drug therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cross-Sectional Cohort: Participants receiving standard of care for hypertension with well-controlled hypertension will participate in 1 visit.
  Interventions: Other: No Intervention
- Longitudinal Cohort: Participants receiving standard of care for hypertension with history of hypertension who are uncontrolled on the current antihypertensive medications or participants with newly diagnosed hypertension (diagnosed within the past 4 weeks and uncontrolled on antihypertensive therapy) will be observed over the course of 12-16 weeks.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention was administered in this study.
  Other Names: No intervention was administered in this study.

SUMMARY:
The purpose of this study is to evaluate blood pressure (BP) goal attainment in adult participants with essential hypertension.

DETAILED DESCRIPTION:
This study has been designed as a non-interventional, observational study to obtain information on hypertension treatment regimens and how well hypertension is controlled in Thai patients in real-life settings. Antihypertensive medications prescribed in this study will be at the discretion of the investigator and the standard of care practice at the particular study site.

The study will enroll approximately 2000 patients. Participants with well-controlled hypertension on their current antihypertensive therapy will participate in the study for only 1 visit. Participants with history of hypertension who are uncontrolled on the current antihypertensive medications or participants with newly diagnosed hypertension (diagnosed within the past 4 weeks and uncontrolled on antihypertensive therapy) will be observed over the course of 12-16 weeks. These participants will make 3 visits to the study site.

This multi-centre trial will be conducted in Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent
2. Age above 18 years.
3. Participants with essential hypertension as per European Society of Hypertension/European Society of Cardiology (ESH/ESC) criteria in general, target blood pressure (BP), systolic blood pressure (SBP) <140 and diastolic blood pressure (DBP) <90 mmHg, in diabetes, target BP, SBP <140 and DBP <85 mmHg, in renal disease with overt proteinuria (urine albumin excretion > 300 mg/day or 200 microgram/min), target BP, SBP <130 and DBP <90 mmHg).

Essential Hypertension will be defined based on the criteria established by the ESH/ESC 2013 criteria:

* Grade 1 Essential hypertension - Systolic blood pressure (SBP) 140 - 159 mmHg and/or diastolic blood pressure (DBP) 90-99 mmHg with no identifiable cause
* Grade 2 Essential hypertension - SBP 160 - 179 mmHg and/or DBP 100 - 109 mmHg with no identifiable cause
* Grade 3 Essential hypertension-SBP ≥ 180 and/or DBP ≥ 110 mmHg with no identifiable cause.

Exclusion Criteria:

1. Female participants who are breastfeeding or pregnant or who are intending to become pregnant.
2. Has known or suspected secondary hypertension.
3. Is currently enrolled in or has not yet completed at least 30 days since ending an investigational product or device study or is receiving other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with essential hypertension will be enrolled from outpatient hospital departments or hospital clinics in Thailand.
Sampling Method: Probability Sample
Enrollment: 2071 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Controlled Treated Hypertension | Up to 16 weeks

SECONDARY OUTCOMES:
Percentage of Participants for Whom Dose of Current Medications was Increased | Up to 16 weeks
Percentage of Participants for Whom Antihypertensive Medications were Switched | Up to 16 weeks
Percentage of Participants for Whom Second Antihypertensive Drug was Added | Up to 16 weeks
Percentage of Participants for Whom One or More of the Compound of Index Treatment was Removed | Up to 16 weeks
Percentage of Participants in Whom There was No Change in Treatment Regimen | Up to 16 weeks
Reason for Choosing the Treatment Regimens in Hypertension Treatment | Up to 16 weeks
Treatment Regimen for Hypertension | Up to 16 weeks
  Treatment regimen for hypertension will be either monotherapy or combination therapy.
Types of Antihypertensive Medications and Medication Classes | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Pathumwan, Bangkok, Thailand